CLINICAL TRIAL: NCT04509180
Title: Comparison of Treatment Outcomes Between Convergent Procedure and Catheter Ablation for Persistent and Longstanding Persistent Atrial Fibrillation
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Lack of funding
Sponsor: University Medical Centre Ljubljana (Other)
Responsible Party: Principal Investigator, Matevz Jan, MD, University Medical Centre Ljubljana
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0120-161/2020/4
Record Dates: First submitted 2020-08-07; First posted 2020-08-11 (Actual); Last update posted 2023-01-18 (Actual); Status verified 2023-01

CONDITIONS: Persistent Atrial Fibrillation; Longstanding Persistent Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation | interventions — Catheter Ablation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Catheter ablation group (Experimental): Patients undergoing catheter procedure will be put under conscious sedation and local anesthesia. Pulmonary vein isolation and posterior wall isolation will be performed with a radiofrequency ablation catheter (20-45W, open-tip irrigation). Ablation index will be used for the lesion formation guidance (450-500 on anterior aspects; 350-400 on the posterior aspects). A wide antral circumferential ablation will be performed for pulmonary veins and a box lesion set for the posterior left atrial wall. Voltage mapping and signal analysis performed by the operator will be used to assess electrical isolation of the pulmonary veins and posterior wall and to identify gaps in ablation lines. At the end of procedure, an implantable loop recorder will be inserted in the left parasternal region.
  Interventions: Procedure: Catheter ablation
- Convergent group (Active Comparator): Patients undergoing convergent procedure will be put under general anesthesia. A minimally invasive epicardial radiofrequency ablation (30W, 90s) of posterior wall will be performed through a subxiphoid window. Monitoring of the esophageal temperature will be performed with an esophageal temperature probe set at 38°C. Next, an endocardial radiofrequency ablation (20-40W, open-tip irrigation; ablation index 450-500 anteriorly and 350-400 posteriorly) of pulmonary veins in a wide antral circumferential fashion will be performed. Voltage mapping and signal analysis performed by the operator will be used to assess the electrical isolation of the pulmonary veins and posterior wall and to identify the gaps in ablation lines. At the end of procedure, an implantable loop recorder will be inserted in the left parasternal region.
  Interventions: Procedure: Convergent procedure

INTERVENTIONS:
Procedure: Catheter ablation — Endovascular approach
  Arms: Catheter ablation group
Procedure: Convergent procedure — Surgical and endovascular approach
  Arms: Convergent group

SUMMARY:
In the last 20 years, atrial fibrillation has become one of the leading healthcare burden in Europe and other developed countries. With an ever-increasing prevalence and incidence, atrial fibrillation is expected to remain a significant problem in the near future. Due to numerous detrimental effects atrial fibrillation has on the patient's health, having an efficient and safe treatment is crucial for managing the problem.

The gold standard for an atrial fibrillation treatment is a catheter ablation. In typical catheter ablation procedure, triggers in pulmonary veins are addressed with a pulmonary vein isolation- offering a high long-term success rate in patients with paroxysmal atrial fibrillation. However, the same cannot be said for persistent and longstanding persistent atrial fibrillation. Studies have shown that efficiency of catheter ablation for persistent and longstanding persistent atrial fibrillation, including multiple procedures per patient, ranges around 50 %. It is postulated that extrapulmonary vein triggers, such as foci located in the posterior wall of the left atrium, play an important role in initiating and maintaining persistent and longstanding persistent atrial fibrillation. In the past, to address this issue, a convergent procedure was developed. In convergent procedure an epicardial ablation of posterior wall is performed through a subxyphoid window. Next, an endocardial ablation with an ablation catheter is performed to isolate pulmonary veins. Because the epicardial lesions are applied in the opposite direction and not towards the esophagus, ablation of posterior wall can safely be performed. The procedure offers a high long-term success rate (85%) in patients with persistent and longstanding persistent atrial fibrillation. However, due to higher associated invasiveness, the convergent procedure carries a higher risk of complications compared with catheter ablation (4 % vs 9 %).

With advancements in ablation catheter technology, such as continuous force measurement at the tip of the catheter, the depth and volume of the lesion can be estimated. This information greatly increases the reliability of lesion formation. The operator can thus effectively apply lesions to the posterior wall of the left atrium more safely in regards to the collateral damage to the esophagus.

The objectives of the study are:

* To compare procedural, safety and efficiency profile of convergent procedure with catheter ablation procedure, both targeting pulmonary veins triggers and triggers located in the posterior wall of the left atrium.
* To compare long-term success rate of convergent procedure with catheter ablation procedure, both targeting pulmonary veins triggers and triggers located in the posterior wall of the left atrium.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed persistent and/or long-term
* Failed medical therapy with antiarrhythmic drug therapy

Exclusion Criteria:

* Expected life expectancy of less than one year
* Previous heart operation
* Previous ablation procedure
* Left ventricular ejection fraction below 30 %
* Severe valvular heart disease
* Acute coronary syndrome
* Diminished functional capacity due to non-cardiac co-morbidities
* Pregnancy

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-02-26 (Actual); Primary Completion 2022-09-01 (Estimated); Study Completion 2024-09-01 (Estimated)

PRIMARY OUTCOMES:
Noninferiority of catheter ablation | 1 year
  arrhythmia-free survival registered with an implantable loop recorder

SECONDARY OUTCOMES:
Differences in AF burden | 1 year
  registered with an implantable loop recorder
Differences in acute success rate of posterior wall isolation | 1 month
  registered with voltage and activation mapping during the index procedure
Differences in complication rate | 1 month
  procedure related complications

CONTACTS AND LOCATIONS:
Locations (1):
- UMC Ljubljana, Ljubljana, Slovenia

IPD SHARING:
Plan to Share IPD: No